CLINICAL TRIAL: NCT06559852
Title: The Impact of Yoga on Endometriosis-Related Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Linda Li, Assistant Professor, Department of Obstetrics and Gynecology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025723
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: Pelvic Pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Intervention (Experimental)
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Participants will engage in a 12-week virtual yoga course to assess impact on endometriosis-related pain

SUMMARY:
The central hypothesis of the investigators is that the practice of yoga will result in an improvement of endometriosis related pain symptoms for women with endometriosis.

DETAILED DESCRIPTION:
Yoga has been demonstrated to improve menstrual pain associated with primary dysmenorrhea through use of physical exercises, mental meditation, and breathing techniques. Still, there has been limited studies assessing potential benefits of yoga on pain symptoms of endometriosis. It is important to further assess yoga as a complementary therapy for women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

1. Reproductive aged women 18-45
2. Self-reported prior surgery with pathology confirming a diagnosis of endometriosis
3. No current use of yoga
4. Baseline moderate pain, score greater than or equal to 5 on VAS scoring
5. Access to internet with wifi capability for zoom platform and completion of weekly surveys
6. Access to items required for yoga session participation (2 blankets or towels, firm pillow, stable chair, wall space, comfortable clothing, water)
7. Ability to commit to duration of 12-week yoga course

Exclusion Criteria:

1. Pregnant patients
2. Established yoga participation or moderate exercise regimen
3. Physical trauma or disability
4. Planned surgery or hormonal medication change during study
5. Non-English speaking patients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Endometriosis Health Profile-30 Pain Score | Baseline to completion at 12-weeks
  Identify the impact of yoga on endometriosis related pain based on the Endometriosis Health Profile-30, with specific focus on the domain of pain. The EHP-30 questionnaire consists of five scales which includes pain, control and powerlessness, emotional well-being, social support, and self-image and a total of 30 questions. Each scale is translated into a score ranging from 0, or the best health status, to 100, the worst health status.

SECONDARY OUTCOMES:
Change in Visual Analog Scale scores | Baseline to completion at 12-weeks
  Comparison of visual analog scale scores from start to the end of the study. The visual analog scale is a validated scale for measuring acute and chronic pain. Scores are recorded on a scale between 0 or "no pain" and 10, the "worst pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish in an ICMJE journal upon completion of study.